CLINICAL TRIAL: NCT07261189
Title: Comparative Study of Staples Versus Polypropylene Sutures for Mesh Fixation in Lichenstein's Tension-free Inguinal Hernia Repair in Terms of Postoperative Pain
Brief Title: Comparing Staples Versus Polypropylene Sutures for Mesh Fixation in Inguinal Hernia Repair in Terms of Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Collaborators: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Asna Ursani, MBBS, FCPS Trainee, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JPMC-GS-2025-12507
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Inguinal Hernia
Keywords: Lichensteins repair; staples; polypropylene sutures; mesh fixation; postoperative pain; hernioplasty
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staples for mesh fixation (Experimental): Mesh secured with stainless steel staples during Lichenstein tension-free inguinal hernioplasty
  Interventions: Procedure: Staples for mesh fixation
- Polypropylene Suture Group (Active Comparator): Mesh secured with polypropylene sutures during Lichensteins tension-free inguinal hernioplasty
  Interventions: Procedure: Polypropylene suture for mesh fixation

INTERVENTIONS:
Procedure: Staples for mesh fixation — Mesh secured using stainless steel staples in Lichenstein tension-free inguinal hernioplasty
  Arms: Staples for mesh fixation
Procedure: Polypropylene suture for mesh fixation — Mesh secured using polypropylene sutures in Lichenstein tension-free inguinal hernioplasty
  Arms: Polypropylene Suture Group

SUMMARY:
This randomized controlled trial aims to compare postoperative pain between staples and polypropylene sutures used for mesh fixation in patients undergoing elective Lichtenstein tension-free inguinal hernia repair.

DETAILED DESCRIPTION:
Inguinal hernia repair is one of the most common general surgical procedures worldwide. The standard method for mesh fixation during Lichtenstein tension-free hernioplasty uses polypropylene sutures. However, skin staples have recently been introduced as a faster and potentially less painful alternative. This randomized controlled trial compares both methods in terms of postoperative pain, measured using the Visual Analogue Scale (VAS), and operative time.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 20 to 60 years.
* Patients undergoing elective Lichtenstein tension-free mesh repair for unilateral, uncomplicated inguinal hernia (direct or indirect).
* Body Mass Index (BMI) between 19 and 30 kg/m².
* ASA physical status I, II, or III.
* Patients willing to participate and provide informed consent.

Exclusion Criteria:

* Diabetic patients (on medical records).
* Bilateral or recurrent inguinal hernia.
* Complicated hernia (irreducible, obstructed, or strangulated).
* Patients unwilling to participate or who fail to complete follow-up.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain (VAS score) | Postoperative day 1, day 7 and day 30
  Pain intensity will be measured using the Visual Analogue Scale (VAS 0-10)

SECONDARY OUTCOMES:
Operative time (minutes) | During Surgery (intraoperative period)
  Time in minutes from initiation of mesh fixation to completion of skin closure

CONTACTS AND LOCATIONS:
Overall Officials: Shafqatullah, Principal Investigator — Jinnah Postgraduate Medical Centre, Karachi, Pakistan
Locations (1):
- Jinnah Postgraduate Medical Centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
This study will not share individual participant data. Only aggregated results will be published. Data will remain confidential as per institutional policy and ethical approval requirements